CLINICAL TRIAL: NCT06788236
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of AVTR101 in Sarcopenia Patients
Brief Title: Study of Efficacy and Safety of AVTR101 in Sarcopenic Elderly
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due subject enrollment delay and to secure expiration of the test drug, it was necessary to minimize the subject enrollment period. In addition, it was deemed advantageous to increase the overall efficiency of the clinical program.
Sponsor: Aventi Biotechnology Inc. (Industry)
Collaborators: Seoul National University Bundang Hospital (Other); Ajou University School of Medicine (Other); SMG-SNU Boramae Medical Center (Other); Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AV-R101-211
Record Dates: First submitted 2024-12-11; First posted 2025-01-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Subjects will take one 120 mg capsule (test drug) three times daily for a total treatment duration of 12 weeks.
  Interventions: Drug: AVTR101
- Placebo Arm (Placebo Comparator): Subjects will take one placebo capsule three times daily for a total treatment duration of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVTR101 — three times daily
  Arms: Treatment Arm
Drug: Placebo — three times daily
  Arms: Placebo Arm

SUMMARY:
The goal of this clinical trial is to primarily evaluate the efficacy of AVTR101 to placebo on physical performance in sarcopenia patients.

Participants will:

Take AVTR101 or a placebo three times daily for 12 weeks Visit the clinic once every 4 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years or older at the time of screening
* Appendicular skeletal muscle mass (ASM) measured by dual-energy x-ray absorptiometry (DXA), men < 7.0 kg/m2, women < 5.4 kg/m2
* Handgrip strength, men < 28 kg, women < 18 kg or 5-times sit-to-stand ≥ 12 second or 6 meter walking speed < 1.0 m/s
* nutrition status confirmed by mini nutritional assessment (MNA) is higher than 8 at the time of screening
* body weight ≥ 35 kg and BMI is between 15~30 kg/m2 at the time of screening
* After fully understanding the written consent, which includes compliance with the requirements and restrictions listed in the trial protocol and describes the overall nature and purpose of the clinical trial, including potential risks and side effects, the subject (or representative) voluntarily A person who signed a written consent form as

Exclusion Criteria:

* Patients with neuromuscular or nervous system diseases (e.g. Parkinson's disease, Lou Gehrig's disease, stroke affecting lower extremity function, muscular dystrophy, epilepsy, multiple sclerosis, etc.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Change in SPPB total score at 12 weeks | From enrollment to the end of treatment at 12 weeks
  The SPPB evaluates lower extremity function through three components: standing balance, usual gait speed, and chair stand. Each component is scored on a scale from 0 to 4, with the total score ranging from 0 to 12. A higher score reflects a higher level of function.

SECONDARY OUTCOMES:
Change in SPPB total score at 4, 8 weeks | From enrollment to the end of treatment at 4, 8 weeks
  The SPPB evaluates lower extremity function through three components: standing balance, usual gait speed, and chair stand. Each component is scored on a scale from 0 to 4, with the total score ranging from 0 to 12. A higher score reflects a higher level of function.
Change in 5-STS time | From enrollment to the end of treatment at 4, 8, 12 weeks
  Change in 5-STS time required at 4, 8, 12 weeks after administration compared to baseline
Change in 6m walk speed | From enrollment to the end of treatment at 4, 8, 12 weeks
  Change in 6m walk speed at 4, 8, 12 weeks after administration compared to baseline
Change in ASM measured by DXA | From enrollment to the end of treatment at 12 weeks
  Change in ASM measured by DXA at 12 weeks after administration compared to baseline
Change in handgrip strength | From enrollment to the end of treatment at 4, 8, 12 weeks
  Change in handgrip strength at 4, 8, 12 weeks after administration compared to baseline
Change in SARC-F total score | From enrollment to the end of treatment at 12 weeks
  The SARC-F is a simple, 5-item screening questionnaire designed to rapidly assess the risk of sarcopenia in older adults. It evaluates five components: Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls. Each item is scored from 0 to 2, resulting in a total score ranging from 0 to 10, with a score of 4 or higher indicating an increased risk of sarcopenia.
Change in SarQoL: total score | From enrollment to the end of treatment at 12 weeks
  The SarQoL (Sarcopenia and Quality of Life) is a validated, sarcopenia-specific quality of life questionnaire designed for older adults. It consists of 22 questions across seven domains: physical and mental health, locomotion, body composition, functionality, activities of daily living, leisure activities, and fears. The questionnaire produces a total score ranging from 0 to 100, with higher scores indicating better quality of life.

OTHER OUTCOMES:
Hematology: RBC | 0, 4, 8, 12 week
  Laboratory test - hematology, Red Blood Cell (10^6/uL)
Hematology: Hemoglobin | 0, 4, 8, 12 week
  Laboratory test - hematology, Hemoglobin (g/dL)
Hematology: Hematocrit | 0, 4, 8, 12 week
  Laboratory test - hematology, Hematocrit (%)
Blood chemistry test: Ca | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, Ca (mg/dL)
Blood chemistry test: ALT | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, ALT (U/L)
Blood chemistry test: AST | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, AST (U/L)
Blood chemistry test: ALP | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, ALP (U/L)
Blood chemistry test: Total bilirubin (mg/dL) | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, Total bilirubin (mg/dL)
Blood chemistry test: γ-GT | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, γ-GT (U/L)
Blood chemistry test: Lactic Dehydrogenase | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, Lactic Dehydrogenase (U/L)
Blood chemistry test: Total Cholesterol | 0, 4, 8, 12 week
  Laboratory tests - Blood chemistry test, Total Cholesterol (mg/dL)
Urinalysis: Leukocyte | 0, 4, 8, 12 week
  Laboratory tests - Urinalysis, Leukocyte (10^2/uL)
Urinalysis: Nitrate | 0, 4, 8, 12 week
  Laboratory tests - Urinalysis, Nitrate (mg/dL)
Electrocardiogram: date and time | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - date and time of ECG
Electrocardiogram: heart rate | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - heart rate (beat per minute, bpm)
Electrocardiogram: PR interval | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - PR interval (millisecond, ms)
Electrocardiogram: QT interval uncorrected | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - QT interval uncorrected (millisecond, ms)
Electrocardiogram: QTc interval | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - QTc interval (millisecond, ms)
Electrocardiogram: QRS duration | 0, 4, 8, 12 week
  12-lead ECG (Electrocardiogram) - QRS duration (millisecond, ms)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University School of Medicine, Suwon, Gyeonggi-do
  - Asan Medical Center, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul